CLINICAL TRIAL: NCT02152865
Title: Clinical Trial of Lupeol for Mild-moderate Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: anti-acne product
Record Dates: First submitted 2014-05-25; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Acne
Keywords: medication
MeSH Terms: conditions — Acne Vulgaris | interventions — lupeol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Lupeol (Active Comparator): Patients are supposed to apply lupeol on one side of face two times per day for 8 weeks
  Interventions: Drug: Lupeol
- Control vehicle (Placebo Comparator): Patients are supposed to apply vehicle control to another side of face two times per day for 8 weeks
  Interventions: Drug: Control vehicle

INTERVENTIONS:
Drug: Lupeol — Patients are supposed to apply lupeol cream to one side of their face two times per day for 8 weeks.
  Other Names: no brand name
  Arms: Lupeol
Drug: Control vehicle — Patients are supposed to apply their control vehicle to the other side of their face for 8 weeks
  Other Names: No brand name
  Arms: Control vehicle

SUMMARY:
For the chemical lupeol isolated from eggplant, we applied it to one side of face, and applied vehicle control to another side for 8 -weeks. The study was performed in a 8-week, randomized controlled, split face fashion. Investigators evaluated safety and efficacy during baseline, 2 weeks, 4weeks, and 8 weeks after beginning of study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age 15 who were clinically diagnosed with mild to moderate acne vulgaris

Exclusion Criteria:

* ; known pregnancy or lactation, any medical illness that might influence the results of the study, a previous history of oral acne medication or surgical procedures including laser treatment within 6 month and topical medication within 4 weeks of study enrollment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Acne lesion counts as a measure of efficacy | 8 weeks after beginning of applications
  Both inflammatory & non-inflammatory acne lesions of both of their facial sides

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks after beggning of applications
  Among total patients enrolled in this study, number of patients either experiencing objective adverse events or subjective uncomfortableness were counted

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea